CLINICAL TRIAL: NCT06903130
Title: An Exploratory, Non-Interventional, Prospective, Multicenter, Nationwide, Clinical Study to Evaluate the Effects of the Complement C5 Inhibitor Ravulizumab on Serum Neurofilament Light Chain (sNfL) and Glial Fibrillary Acidic Protein (sGFAP) Levels in Patients With Aquaporin-4-Positive (AQP4-Ab+) Neuromyelitis Optica Spectrum Disorder (NMOSD)
Brief Title: Clinical Study to Evaluate the Effects of the Complement C5 Inhibitor Ravulizumab on Serum Neurofilament Light Chain (sNfL) and Glial Fibrillary Acidic Protein (sGFAP) Levels in Patients With Aquaporin-4-Positive (AQP4-Ab+) Neuromyelitis Optica Spectrum Disorder (NMOSD)
Status: Not yet recruiting | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Georgios Tsivgoulis, Professor & Chairman of Second Department of Neurology, School of Medicine, National & Kapodistrian University of Athens, "Attikon" University Hospital, Athens, Greece, National and Kapodistrian University of Athens
Other Study IDs: ESR-24-22351
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: NMOSD
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples Without DNA — Serum samples for sNfL and sGFAP levels
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AQP4-IgG seropositive NMOSD patients receiving complement inhibitor treatment: AQP4-IgG seropositive NMOSD patients receiving complement inhibitor treatment with Ravulizumab (group A)
  Interventions: Diagnostic Test: Blood samples for sNfL and sGFAP levels
- AQP4-IgG seropositive NMOSD patients receiving off-label ISTs: AQP4-IgG seropositive NMOSD patients receiving off-label ISTs including rituximab, corticosteroids, azathioprine, and mycophenolate mofetil (group B)
  Interventions: Diagnostic Test: Blood samples for sNfL and sGFAP levels

INTERVENTIONS:
Diagnostic Test: Blood samples for sNfL and sGFAP levels — Blood samples for sNfL and sGFAP levels

SUMMARY:
This is a nationwide observational study looking at how ravulizumab, a complement C5 inhibitor, affects blood biomarkers o sNfL and sGFAP in people with AQP4-antibody positive NMOSD. The study does not change your treatment-only regular blood samples are collected to monitor these markers

DETAILED DESCRIPTION:
This is an exploratory, non-interventional, prospective, multicenter, clinical study. The maximum total number of 40 patients with a diagnosis of seropositive AQP4-IgG NMOSD is expected to be enrolled. The goal is to include at least one-third of these patients in the complement inhibitor ravulizumab group, with the remaining patients in the off-label ISTs group based on current therapeutic clinical practice in Greece. Multiple Neurological Departments with experience in NMOSD diagnosis and treatment will participate. Eligible patients will be recruited in both groups and each participant will be followed up approximately every 60 days for 24 months.

Data Source(s):

Study-related data will be collected and recorded at specific and predetermined data collection timepoints, during routine clinical and laboratory assessments. Information related to the patients' medical history will be collected for the NMOSD patients from each neurological department's database (records/files/electronic database) and patient self-reports. Baseline characteristics (age, sex, height, body weight, and BMI) will also be recorded for all participants.

Study Population:

The target population in the study will include diagnosed patients with AQP4-IgG seropositive NMOSD. Age ≥ 18 years with a history of ≥ 1 NMOSD clinical attack according to 2015 NMOSD criteria. The participants should be undergoing treatment either with off-label ISTs (corticosteroids, azathioprine, mycophenolate mofetil, rituximab) or complement inhibitor therapy with ravulizumab. Corticosteroids can be used as add-on therapy to ravulizumab or the off-label ISTs

Procedures:

1. Measurement of sNfL levels.
2. Measurement of sGFAP levels.
3. Clinical assessment: neurological examination/disability evaluation based on the EDSS.
4. Brain/spinal cord MRI: the number, size, anatomical location of lesions will be assessed. Gadolinium enhancement will also be evaluated whenever post-gadolinium T1-weighted MRI images are available.

   * Scheduled serum collection time points for biomarker measurements (sGFAP, sNfL) and clinical assessments: at the first data recording at Visit 1 and subsequently every 60 (±15) days during the follow-up period, which is set at 24 months.
   * Interim timepoints related to clinical episodes for serum collection of biomarker measurements (sGFAP, sNfL) and clinical assessments: at the onset of a clinical episode (48-hours window).
   * All participants will be clinically evaluated during scheduled follow-ups for sample acquisition or during attack-related visits; clinical evaluation will include neurological examination, MRI evaluation whenever applicable, clinical disability assessment by the EDSS and routine blood test assessment.

ELIGIBILITY:
Inclusion Criteria

Patients are eligible to be included in the study only if all of the following criteria apply:

Age

1. Patient must be 18 years of age or older, at the time of signing the informed consent.

   Type of Patient and Disease Characteristics
2. Anti-AQP4 Ab-positive at screening and a diagnosis of NMOSD as defined by the 2015 international consensus diagnostic criteria (Wingerchuk, 2015). A historically positive anti-AQP4 Ab test may be acceptable if the test was performed using an acceptable, validated cell-based assay from an accredited laboratory.
3. At least 1 clinical attack prior to the Prescreening/Screening Periods.
4. Treatment-naïve patients or patients under specific off-label treatments (rituximab, corticosteroids, azathioprine, mycophenolate mofetil) or the complement C5 inhibitor ravulizumab. Naïve patients who initiate ravulizumab at enrolment, should have been prescribed ravulizumab, but not yet initiated treatment, according to the label and local market reimbursement criteria.
5. Vaccinated against N. meningitidis (for serogroups A, C, W, Y and B) a) within 3 years and at least 2 weeks prior to the first dose of ravulizumab, or b) at the time of the first dose of ravulizumab provided that antibacterial drug prophylaxis is administered as per National Vaccination Guidelines and Summary of Product Characteristics of ravulizumab.

   Weight
6. Body weight ≥ 40 kg.

   Sex
7. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those receiving each immunotherapy.

   Informed Consent
8. Capable of giving signed informed consent as described in Section 10.1.3, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria

Patients are excluded from the study if any of the following criteria apply:

Medical Conditions

1. History of N. meningitidis infection.
2. Human immunodeficiency virus (HIV) infection (evidenced by HIV-1 or HIV-2 antibody titer)
3. History of unexplained infections.
4. Active systemic bacterial, viral, or fungal infection within 14 days prior to screening.
5. Presence of fever ≥ 38°C (100.4°F) within 7 days prior to screening
6. NMOSD pregnant women will be excluded according to the local clinical practice. '
7. History of implanted medical devices which are incompatible with strong magnetic fields used for MRI.

Prior/Concomitant Therapy 6. Use of inebilizumab within 6 months prior to Enrollment in patients switching to another therapy i.e. ravulizumab or the off-label ISTs.

7. Use of satralizumab within 3 months prior to Enrollment. 8. Pregnant, breastfeeding, or intending to conceive during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population in the study will include diagnosed patients with AQP4-IgG seropositive NMOSD. Age ≥ 18 years with a history of ≥ 1 NMOSD clinical attack according to 2015 NMOSD criteria1. The participants should be undergoing treatment either with off-label ISTs (corticosteroids, azathioprine, mycophenolate mofetil, rituximab) or complement inhibitor therapy with ravulizumab. Corticosteroids can be used as add-on therapy to ravulizumab or the off-label ISTs.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
• Changes in sNfL and sGFAP levels during disease course in AQP4-IgG NMOSD seropositive patients receiving Ravulizumab | 2 years
  To evaluate sNfL and sGFAP levels and their fluctuations over time in AQP4-IgG seropositive NMOSD patients receiving complement inhibitor Ravulizumab

SECONDARY OUTCOMES:
Correlation analysis of sGFAP and sNfL levels with the EDSS score. | 2 years
  To evaluate the association of sGFAP and sNfL levels with clinical disability.

OTHER OUTCOMES:
Changes in sGFAP levels in patients experiencing relapse | 2 years
  To assess the clinical utility of sGFAP levels in AQP4-IgG seropositive NMOSD patients to predict clinical relapse risk.
Alterations in sNfL and sGFAP levels during disease course in AQP4-IgG NMOSD seropositive patients receiving receiving off-label ISTs | 2 years
  To investigate for alterations in sNfL and sGFAP levels over time in AQP4-IgG seropositive NMOSD patients receiving off-label ISTs

CONTACTS AND LOCATIONS:
Locations (1):
- Second Department of Neurology, "Attikon" University Hospital, School of Medicine, National and Kapodistrian University of Athens, Athens, Greece